CLINICAL TRIAL: NCT06443710
Title: A Phase I Clinical Study of the Pharmacokinetics and Safety of Technetium [99mTc]-H7ND Injection in Patients With Gastrointestinal Malignancies and Healthy Volunteers
Brief Title: Technetium [99mTc]-H7ND in Patients With Gastrointestinal Malignancies and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiaxing Pharmadax Genesis Pharmaceutical Technology Co.,Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023LP02630
Record Dates: First submitted 2024-05-23; First posted 2024-06-05 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Technetium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with malignant tumors of the gastrointestinal tract or healthy subjects (Experimental): Each patient will receive 10 or 20 mCi ± 20% technetium [99mTc]-H7ND injection intravenously
  Interventions: Drug: Technetium [99mTc]-H7ND injection

INTERVENTIONS:
Drug: Technetium [99mTc]-H7ND injection — Technetium [99mTc]-H7ND injection is a radiolabeled fibroblast activation protein inhibitor

SUMMARY:
The primary objective of this study is: to evaluate the safety of technetium [99mTc]-H7ND injection in patients with gastrointestinal malignancies and in healthy subjects. The secondary objectives of this study are: (1) to examine the pharmacokinetics of technetium [99mTc]-H7ND Injection in healthy subjects. (2) Detect the metabolic stability of technetium [99mTc]-H7ND injection in healthy humans. (3) Detect the biodistribution and estimate the absorbed dose of radiation from internal irradiation of technetium [99mTc]-H7ND injection in patients with malignant tumors of the gastrointestinal tract and in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects should be adult males or females aged 18-75 years (including borderline values, based on the time of signing the informed consent form) at screening, and not less than 1/3 of the total number of cases of each gender
2. All subjects who are males or females of childbearing potential must be using effective contraception during the study period (effective contraception means sterilization, intrauterine hormonal devices, condoms, contraceptive pills/agents, abstinence, or vasectomy)
3. All subjects are fully aware of the purpose, nature, methods, and possible adverse effects of the trial, voluntarily participate and sign a written informed consent form, and are able to follow the protocol requirements to complete the study
4. Healthy subjects with a body mass index within the range of 18.0 to 26.0 kg/m2 (including the borderline value), male subjects weighing ≥ 50 kg, female subjects weighing ≥ 45 kg
5. Healthy subjects are in good health or do not have a history of major diseases
6. Vital signs, physical examination, laboratory tests, and 12-lead electrocardiogram (ECG) results of healthy subjects during the screening period are not abnormal or the abnormalities are not clinically significant.
7. Gastrointestinal malignant tumor subjects with histologically/cytologically confirmed diagnosis of gastrointestinal malignant tumors (including stomach, small intestine and colorectum)
8. Subjects with gastrointestinal malignant tumors with an ECOG score of 0 - 1
9. Subjects with gastrointestinal malignant tumors Blood routine: WBC ≥ 3 × 109 / L, ANC ≥ 1.5 × 109 / L, Hb ≥ 90 g / L, PLT ≥ 75 × 109 / L; Liver function: TBIL ≤ 1.5 × ULN, ALT, AST ≤ 3 × ULN (≤ 5 × ULN for liver metastases); Kidney function: Cr ≤ 1.5 × ULN; Coagulation function: Prothrombin time (PT) ≤1.5×ULN, activated partial thromboplastin time (APTT) ≤1.5×ULN, international normalized ratio (INR) ≤1.5×ULN; Electrolytes: corrected magnesium ≥LLN, allowed to correct electrolytes during the screening period Cardiac function: left ventricular ejection fraction ≥ 50%
10. Subjects who have recovered to Grade 1 (CTCAE Version 5.0) from damage caused by other therapies, except: alopecia, hyperpigmentation; and if nutritionally stable, the presence of irrecoverable long-term toxicity as determined by the Investigator is permitted.
11. Subjects with gastrointestinal malignancies expected to survive ≥ 12 weeks

Exclusion Criteria:

1. Pregnant (positive screening pregnancy test) or breastfeeding female
2. History of alcohol or drug abuse/dependence
3. Known allergy to radioactive rays, or history of other severe allergies
4. Human immunodeficiency virus (HIV) positive or not definitively negative, hepatitis C virus (HCV) or syphilis spirochete antibody test positive, hepatitis B virus (HBV) surface antigen positive and quantitative HBV DNA test ≥ 1.0×103 IU/mL
5. Significant occupational exposure to ionizing radiation in the past 10 years
6. Unable to repeat venipuncture
7. Participation in a clinical study of another drug within 30 days prior to screening and use of another test drug
8. Other conditions that, in the opinion of the investigator, make participation in this clinical trial inappropriate
9. Subjects with gastrointestinal malignancies requiring treatment of symptomatic brain metastases
10. Subjects with gastrointestinal malignancies who have a history of other malignancies, except for malignant lesions that have been treated with therapeutic measures 5 or more years prior to the initiation of investigational drug use and are not known to be active, and who, in the judgment of the Investigator, are at low risk of recurrence. Adequately treated non-melanoma skin cancer or malignant freckle-like nevus without evidence of disease progression. Adequately treated in situ cervical cancer with no evidence of progression. Intraepithelial tumor of the prostate gland without evidence of prostate adenocarcinoma
11. Subjects with gastrointestinal malignancies who have developed clinically significant cardiovascular disease (including, but not limited to, myocardial infarction, unstable angina pectoris, symptomatic congestive heart failure, and uncontrolled severe arrhythmia) within 6 months prior to initiation of study drug use
12. Subjects with gastrointestinal malignancies who have hypertension that is uncontrollable with a single agent
13. Subjects with malignant tumors of the gastrointestinal tract who have a history of hepatic disease or other conditions that interfere with the absorption, distribution, excretion, or metabolism of the drug, as determined by the investigator
14. Subjects with gastrointestinal malignancies have a history of coagulopathy or coagulation disorders.
15. History of arterial or venous embolism in subjects with gastrointestinal malignancies
16. Subjects with gastrointestinal malignancies who, in the judgment of the investigator, have received any medications and treatments prior to enrollment that may interfere with the trial data or that may have resulted in serious side effects that have not been fully cleared
17. Subjects with gastrointestinal malignancies who have an active or uncontrolled infection requiring systemic therapy within 14 days prior to initiation of study drug use
18. Subjects with malignant tumors of the gastrointestinal tract who have undergone major surgical procedures within 28 days prior to the start of investigational drug use-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Security Indicators | 1-7 days from time of injection
  Evaluation of adverse events and serious adverse events according to the Common Terminology Criteria for the Evaluation of Adverse Events (NCI-CTCAE) version 5.0

SECONDARY OUTCOMES:
uptake value ratio | 3 days after injection
  Measure the count ratio of technetium [99mTc]-H7ND tumor area to blood pool, surrounding normal tissue, liver, and muscle in the integrated region of interest.
biodiversity distribution | 3 days after injection
  SPECT/CT whole-body scans were performed at different time points after drug injection to obtain radioactivity counts (%ID) in each major irradiated organ at each time phase to reflect the biodistribution of the drug in the body
internal radiation dose | 3 days after injection
  Plot the "time-activity count" curve for each major organ and calculate the area under the curve. Calculate the retention time of each major exposed organ and apply the software to estimate the absorbed dose of internal radiation for each major exposed organ.
Concentration of technetium [99mTc] H7ND prototype and its radioactive metabolites | Predose and up to 72 hours postdose
  Blood samples were collected at different time points after drug injection, and urine samples were collected at different time intervals for detection of technetium [99mTc] H7ND prototype and its radioactive metabolites using either a radioactive HPLC detector or a radioactive TLC detector.
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  Cmax
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  AUC(0-t)
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  AUC(0-∞)
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  Tmax
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  T1/2
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  AUC_%Extrap
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  CL
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  Vd
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  MRT
Pharmacokinetic parameters | Predose and up to 72 hours postdose
  λz

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No